CLINICAL TRIAL: NCT05775809
Title: Prospective Clinical Cohort Study of Depression
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Yanhui Liao, Major Investigators, Sir Run Run Shaw Hospital
Other Study IDs: 2022-0334
Record Dates: First submitted 2023-02-10; First posted 2023-03-20 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Selective Serotonin Reuptake Inhibitors; Psychotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Patients with major depressive disorder: We collect data of patients with major depressive disorder at different point (baseline, 2nd weekend±7days, 6th weekend±14days, 8th weekend±14days, 12th weekend±14days, Week 14-104 Every 4 weekends ± 14 days).
  Interventions: Drug: selective serotonin reuptake inhibitors; Device: TMS

INTERVENTIONS:
Drug: selective serotonin reuptake inhibitors — Research Treatment Drug treatment The patient did not take antidepressant treatment at least 14 days before enrollment (the patients treated with fluoxetine before enrollment should stop using it for at least 28 days). During 8 weeks, all subjects with major depressive disorder received effective dosages of selective serotonin reuptake inhibitors, and all subjects with major depressive disorder were limited to a single class of antidepressants. If the treatment of selective serotonin reuptake inhibitors is not effective after eight weeks, the drugs can be considered for replacement. The drugs for replacement include but are not limited to selective serotonin reuptake inhibitors.
  Other treatment Settings Psychotherapy and TMS are allowed. The method, frequency, and duration of therapy should be recorded.
  Other Names: Psychotherapy and TMS
Device: TMS — TMS are allowed. The method, frequency, and duration of therapy should be recorded.

SUMMARY:
This is a prospective clinical cohort study of depression. The study was intended to include 300 patients with depression and 100 healthy controls. The study consisted of two phases: the baseline period and the follow-up period, in which all subjects were comprehensively collected, and the follow-up period in which all subjects were followed up at least once a year and data were collected. For patients with major depressive disorder, the follow-up methods included fixed visit and planned visit, and the follow-up time point covered the whole course of depressive disease(baseline, 2nd weekend±7days, 6th weekend±14days, 8th weekend±14days, 12th weekend±14days, Week 14-104 Every 4 weekends ± 14 days). Based on standardized, multi-strategy follow-up system and mobile health technology, long-term follow-up of patients with major depressive disorder was realized, and key nodes of patients' disease fluctuations were captured in time. High quality multidimensional data were collected, including demographic, clinical, EEG and eye movement data. Finally, the objective index system of depression was constructed, and the diagnosis, efficacy/recurrence prediction and suicide warning models of depression were established.

DETAILED DESCRIPTION:
1. Research Treatment

   1.1 Drug treatment

   The patient did not take antidepressant treatment at least 14 days before enrollment (the patients treated with fluoxetine before enrollment should stop using it for at least 28 days). During 8 weeks, all subjects with major depressive disorder received effective dosages of selective serotonin reuptake inhibitors, and all subjects with major depressive disorder were limited to a single class of antidepressants. If the antidepressant treatment plan needed to be adjusted, one antidepressant should be selected as far as possible, and combined treatment with two or more antidepressants should not be allowed. Antipsychotics and mood stabilizers are not permitted. If the treatment of selective serotonin reuptake inhibitors is not effective after eight weeks, the drugs can be considered for replacement. The drugs for replacement include but are not limited to selective serotonin reuptake inhibitors.

   1.2 Other treatment Settings

   Psychotherapy and TMS are allowed. The method, frequency, and duration of therapy should be recorded.

   1.3 Treatment compliance

   Participants were reminded to follow the medication regimen and their medication use was recorded at each visit. Non-use of prescription drugs for ≥70% of the time is considered noncompliance, and the reason for noncompliance should be checked. If there was a protocol violation, the protocol violation was recorded and the follow-up was continued as scheduled.
2. Observation index

Main observation indicators:

Clinical effect: Changes of clinical symptoms in acute phase, maintenance phase and long-term follow-up period. Changes in HAMD-17 scores at different follow-up points compared with baseline were used as the main efficacy evaluation index in this study. The evaluation criteria of clinical efficacy and significant endpoints at different stages are as follows:

① Early onset: The total score of HAMD-17 decreased by more than 20% from baseline after 2 weeks of treatment;

② Effective: The total score of HAMD-17 was reduced by more than 50% compared with baseline; Stable and effective was defined as two consecutive HAMD-17 scores decreased by more than 50% from baseline at the 8th weekend of the acute phase.

2.1 A method of measuring or evaluating observational indicators

1) General demographic data survey The patient's date of birth, gender, height, weight, nationality, marital status, occupation type and years of education were investigated.

Clinical information collection

2）Medical history information:

* Time of first onset of major depressive disorder/bipolar disorder
* The onset of the current depressive episode
* Total episodes (including this one) : depressive episodes

2.2 Scale evaluation(baseline, 2nd weekend±7days, 6th weekend±14days, 8th weekend±14days, 12th weekend±14days, Week 14-104 Every 4 weekends ± 14 days)：

We collect scale data of patients with major depressive disorder at different point (baseline, 2nd weekend±7days, 6th weekend±14days, 8th weekend±14days, 12th weekend±14days, Week 14-104 Every 4 weekends ± 14 days), and collect scale data of healthy controls during the baseline period.

self-rating scale： Snaith-Hamilton Pleasure Scale, SHAPS Generalized Anxiety Disorder,GAD-7 Patient Health Questionnare, PHQ-9 Hypomania Check List,HCL-33 Sheehan Disability Scale，SDS Childhood Trauma Questionnaire，CTQ Big 5 Personality Questionnaire， B5PQ Dysfunctional Attitude Scale，DAS Interpersonal Reactivity Index-C Scale for Suicide Ideation，SSI

Other rating scale Hamilton Depression Rating Scale for Depression - 17-item，HAMD-17 Hamilton Anxiety Scale，HAMA Brief Psychiatric Rating Scale, BPRS 4 items

2.3 EEG and eye movement data collection (baseline, 2nd weekend±7days, 6th weekend±14days, 8th weekend±14days, 12th weekend±14days, Week 14-104 Every 4 weekends ± 14 days)

We collect EEG and eye movement data of patients with major depressive disorder at different point(baseline, 2nd weekend±7days, 6th weekend±14days, 8th weekend±14days, 12th weekend±14days, Week 14-104 Every 4 weekends ± 14 days), and collect EEG and eye movement data of healthy controls during the baseline period.

ELIGIBILITY:
Inclusion Criteria:

* Out-patient or in-patient aged 18-65 years (including 18 and 65 years), regardless of gender;
* The Chinese version of the Concise International Neuropsychiatric Interview (M.I.N.I.) 7.0.2 type interview, in line with the DSM-5 Diagnostic criteria for major depressive disorder, either first or recurrent;
* Screening and baseline Hamilton Depression Scale (HAMD-17) Score ≥14;
* No antidepressants were taken for at least 14 days prior to enrollment (patients treated with fluoxetine prior to enrollment should Stop for at least 28 days);
* A single class of antidepressant medication is planned;
* Primary school education or above, able to understand the research content;
* Understand and voluntarily participate in this study, and I sign the informed consent.

Exclusion Criteria:

* A current or previous DSM-5 diagnosis of a major mental disorder other than major depressive disorder, Such as neurodevelopmental disorders, neurocognitive disorders, schizophrenia and other psychotic disorders, bipolar disorder Sensory disorder, obsessive disorder, panic disorder, post-traumatic stress disorder, alcohol (or drug) dependence or abuse User and personality disorder;
* depression secondary to an organic mental disorder caused by a systemic disease or a neurological disease Seizures, such as depression caused by hypothyroidism;
* Severe or unstable cardiovascular, respiratory, liver, kidney, endocrine, hematological or other conditions Other systemic diseases were not considered suitable for inclusion in this study.
* During the screening period or baseline period, the investigators considered that the physical examination and laboratory examination of the patients were abnormal and judged to have significant clinical significance Bedsense;
* had received systemic Modified Electric therapy (Modified Electric) 3 months before screening Convulsive Therapy, MECT) or Transcranial Magnetic stimulation (Transcranial Magnetic Stimulation (TMS), Deep Brain Stimulation (DBS), Vagus Nerve Stimulation (VNS);
* The withdrawal of psychotropic drugs did not reach 7 half-lives before screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Depression is a mental state characterized by persistent low mood, loss of interest and pleasure in daily activities, autonomic disorders and decreased energy, resulting in varying degrees of impairment of social and occupational functioning.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-05-20 (Estimated)

PRIMARY OUTCOMES:
score of Snaith-Hamilton Pleasure Scale, SHAPS | baseline
  rating scale
Generalized Anxiety Disorder,GAD-7 | baseline
  rating scale
Patient Health Questionnare, PHQ-9 | baseline
  rating scale
Hypomania Check List,HCL-33 | baseline
  rating scale
Sheehan Disability Scale，SDS | baseline
  rating scale
Childhood Trauma Questionnaire，CTQ | baseline
  rating scale
Big 5 Personality Questionnaire， B5PQ | baseline
  rating scale
Dysfunctional Attitude Scale，DAS | baseline
  rating scale
Interpersonal Reactivity Index-C | baseline
  rating scale
Scale for Suicide Ideation，SSI | baseline
  rating scale
Hamilton Depression Rating Scale for Depression - 17-item，HAMD-17 | baseline
  rating scale
Hamilton Anxiety Scale，HAMA | baseline
  rating scale
Brief Psychiatric Rating Scale, BPRS 4 items | baseline
  rating scale
score of Snaith-Hamilton Pleasure Scale, SHAPS | 2nd weekend±7days,
  rating scale
score of Generalized Anxiety Disorder,GAD-7 | 2nd weekend±7days,
  rating scale
score of Patient Health Questionnare, PHQ-9 | 2nd weekend±7days,
  rating scale
score of Hypomania Check List,HCL-33 | 2nd weekend±7days,
  rating scale
score of Sheehan Disability Scale，SDS | 2nd weekend±7days,
  rating scale
score of Interpersonal Reactivity Index-C | 2nd weekend±7days,
  rating scale
score of Scale for Suicide Ideation，SSI | 2nd weekend±7days,
  rating scale
Hamilton Depression Rating Scale for Depression - 17-item，HAMD-17 | 2nd weekend±7days,
  rating scale
Hamilton Anxiety Scale，HAMA | 2nd weekend±7days,
  rating scale
score of Snaith-Hamilton Pleasure Scale, SHAPS | 6th weekend±14days,
  rating scale
Generalized Anxiety Disorder,GAD-7 | 6th weekend±14days,
  rating scale
Patient Health Questionnare, PHQ-9 | 6th weekend±14days,
  rating scale
Hypomania Check List,HCL-33 | 6th weekend±14days,
  rating scale
Sheehan Disability Scale，SDS | 6th weekend±14days,
  rating scale
Interpersonal Reactivity Index-C | 6th weekend±14days,
  rating scale
Scale for Suicide Ideation，SSI | 6th weekend±14days,
  rating scale
Hamilton Depression Rating Scale for Depression - 17-item，HAMD-17 | 6th weekend±14days,
  rating scale
Hamilton Anxiety Scale，HAMA | 6th weekend±14days,
  rating scale
score of Snaith-Hamilton Pleasure Scale, SHAPS | 8th weekend±14days,
  rating scale
score of Generalized Anxiety Disorder,GAD-7 | 8th weekend±14days,
  rating scale
score of Patient Health Questionnare, PHQ-9 | 8th weekend±14days,
  rating scale
score of Hypomania Check List,HCL-33 | 8th weekend±14days,
  rating scale
score of Sheehan Disability Scale，SDS | 8th weekend±14days,
  rating scale
score of Interpersonal Reactivity Index-C | 8th weekend±14days,
  rating scale
score of Scale for Suicide Ideation，SSI | 8th weekend±14days,
  rating scale
score of Hamilton Depression Rating Scale for Depression - 17-item，HAMD-17 | 8th weekend±14days,
  rating scale
score of Hamilton Anxiety Scale，HAMA | 8th weekend±14days,
  rating scale
score of Snaith-Hamilton Pleasure Scale, SHAPS | 12th weekend±14days,
  rating scale
score of Generalized Anxiety Disorder,GAD-7 | 12th weekend±14days,
  rating scale
score of Patient Health Questionnare, PHQ-9 | 12th weekend±14days,
  rating scale
score of Hypomania Check List,HCL-33 | 12th weekend±14days,
  rating scale
score of Sheehan Disability Scale，SDS | 12th weekend±14days,
  rating scale
score of Interpersonal Reactivity Index-C | 12th weekend±14days,
  rating scale
score of Scale for Suicide Ideation，SSI | 12th weekend±14days,
  rating scale
score of Hamilton Depression Rating Scale for Depression - 17-item，HAMD-17 | 12th weekend±14days,
  rating scale
score of Hamilton Anxiety Scale，HAMA | 12th weekend±14days,
  rating scale
score of Snaith-Hamilton Pleasure Scale, SHAPS | Week 14-104 Every 4 weekends ± 14 days
  rating scale
Generalized Anxiety Disorder,GAD-7 | Week 14-104 Every 4 weekends ± 14 days
  rating scale
score of Patient Health Questionnare, PHQ-9 | Week 14-104 Every 4 weekends ± 14 days
  rating scale
score of Hypomania Check List,HCL-33 | Week 14-104 Every 4 weekends ± 14 days
  rating scale
score of Sheehan Disability Scale，SDS | Week 14-104 Every 4 weekends ± 14 days
  rating scale
score of Interpersonal Reactivity Index-C | Week 14-104 Every 4 weekends ± 14 days
  rating scale
score of Scale for Suicide Ideation，SSI | Week 14-104 Every 4 weekends ± 14 days
  rating scale
score of Hamilton Depression Rating Scale for Depression - 17-item，HAMD-17 | Week 14-104 Every 4 weekends ± 14 days
  rating scale
score of Hamilton Anxiety Scale，HAMA | Week 14-104 Every 4 weekends ± 14 days
  rating scale
average power of 4 bands: δ (1-4 Hz)、 θ (4-8 Hz)、 α (8-13 Hz)、 β (13-30 Hz) | baseline
  EEG features
1.Average duration of EEG microstates 2. The average number of occurrences of EEG microstates per second 3. Average percentage of time covered by EEG microstates 4.the calculation of microstate transition. | baseline
  EEG features
Connectivity index of full-band brain function network, and connectivity index of each band brain function network | baseline
  EEG features
EEG features extracted by machine learning | baseline
  EEG features
average power of 4 bands: δ (1-4 Hz)、 θ (4-8 Hz)、 α (8-13 Hz)、 β (13-30 Hz) | 2nd weekend±7days
  EEG features
Average duration of EEG microstates 2. The average number of occurrences of EEG microstates per second 3. Average percentage of time covered by EEG microstates 4.the calculation of microstate transition. | 2nd weekend±7days
  EEG features
Connectivity index of full-band brain function network, and connectivity index of each band brain function network | 2nd weekend±7days
  EEG features
EEG features extracted by machine learning | 2nd weekend±7days
  EEG features
average power of 4 bands: δ (1-4 Hz)、 θ (4-8 Hz)、 α (8-13 Hz)、 β (13-30 Hz) | 6th weekend±14days
  EEG features
1.Average duration of EEG microstates 2. The average number of occurrences of EEG microstates per second 3. Average percentage of time covered by EEG microstates 4.the calculation of microstate transition. | 6th weekend±14days
  EEG features
Connectivity index of full-band brain function network, and connectivity index of each band brain function network | 6th weekend±14days
  EEG features
EEG features extracted by machine learning | 6th weekend±14days
  EEG features
average power of 4 bands: δ (1-4 Hz)、 θ (4-8 Hz)、 α (8-13 Hz)、 β (13-30 Hz) | 8th weekend±14days
  EEG features
1.Average duration of EEG microstates 2. The average number of occurrences of EEG microstates per second 3. Average percentage of time covered by EEG microstates 4.the calculation of microstate transition. | 8th weekend±14days
  EEG features
Connectivity index of full-band brain function network, and connectivity index of each band brain function network | 8th weekend±14days
  EEG features
EEG features extracted by machine learning | 8th weekend±14days
  EEG features
average power of 4 bands: δ (1-4 Hz)、 θ (4-8 Hz)、 α (8-13 Hz)、 β (13-30 Hz) | 12th weekend±14days
  EEG features
1.Average duration of EEG microstates 2. The average number of occurrences of EEG microstates per second 3. Average percentage of time covered by EEG microstates 4.the calculation of microstate transition. | 12th weekend±14days
  EEG features
Connectivity index of full-band brain function network, and connectivity index of each band brain function network | 12th weekend±14days
  EEG features
EEG features extracted by machine learning | 12th weekend±14days
  EEG features
average power of 4 bands: δ (1-4 Hz)、 θ (4-8 Hz)、 α (8-13 Hz)、 β (13-30 Hz) | Week 14-104 Every 4 weekends ± 14 days
  EEG features
1.Average duration of EEG microstates 2. The average number of occurrences of EEG microstates per second 3. Average percentage of time covered by EEG microstates 4.the calculation of microstate transition. | Week 14-104 Every 4 weekends ± 14 days
  EEG features
Connectivity index of full-band brain function network, and connectivity index of each band brain function network | Week 14-104 Every 4 weekends ± 14 days
  EEG features
EEG features extracted by machine learning | Week 14-104 Every 4 weekends ± 14 days
  EEG features
Eye movement index | baseline
  Collect resting eye movement data and task eye movement data. For eye movement data, features are extracted from blinking, scanning, staring, pupil diameter, initial fixation latency, initial fixation duration, total fixation duration and area of interest and so on.
Eye movement index | 2nd weekend±7days
  Collect resting eye movement data and task eye movement data. For eye movement data, features are extracted from blinking, scanning, staring, pupil diameter, initial fixation latency, initial fixation duration, total fixation duration and area of interest and so on.
Eye movement index | 6th weekend±14days
  Collect resting eye movement data and task eye movement data. For eye movement data, features are extracted from blinking, scanning, staring, pupil diameter, initial fixation latency, initial fixation duration, total fixation duration and area of interest and so on.
Eye movement index | 8th weekend±14days
  Collect resting eye movement data and task eye movement data. For eye movement data, features are extracted from blinking, scanning, staring, pupil diameter, initial fixation latency, initial fixation duration, total fixation duration and area of interest and so on.
Eye movement index | 12th weekend±14days
  Collect resting eye movement data and task eye movement data. For eye movement data, features are extracted from blinking, scanning, staring, pupil diameter, initial fixation latency, initial fixation duration, total fixation duration and area of interest and so on.
Eye movement index | Week 14-104 Every 4 weekends ± 14 days
  Collect resting eye movement data and task eye movement data. For eye movement data, features are extracted from blinking, scanning, staring, pupil diameter, initial fixation latency, initial fixation duration, total fixation duration and area of interest and so on.
Eye movement features extracted by machine learning | baseline
  Eye movement features extracted by machine learning
Eye movement features extracted by machine learning | 2nd weekend±7days
  Eye movement features extracted by machine learning
Eye movement features extracted by machine learning | 6th weekend±14days
  Eye movement features extracted by machine learning
Eye movement features extracted by machine learning | 8th weekend±14days
  Eye movement features extracted by machine learning
Eye movement features extracted by machine learning | 12th weekend±14days
  Eye movement features extracted by machine learning
Eye movement features extracted by machine learning | Week 14-104 Every 4 weekends ± 14 days
  Eye movement features extracted by machine learning

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China